CLINICAL TRIAL: NCT02514408
Title: The Impact Radical Cystectomy Has on the Expulsion of Circulating Tumor Cells
Brief Title: Circulating Tumor Cells in Operative Blood in Patients With Bladder Cancer
Status: Withdrawn | Type: Observational
Why Stopped: No funding
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 4B-15-7; NCI-2015-01063 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 4B-15-7 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2015-07-30; First posted 2015-08-03 (Estimated); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Stage II Bladder Urothelial Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (collection of blood samples): Patients undergo placement of a central line via the right femoral vein and undergo ORC. Blood samples are collected and analyzed for CTCs pre-surgery, at 30 minutes and 1 hour once ORC begins, post-surgery, and 7 days after surgery.
  Interventions: Procedure: Catheter Management; Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Catheter Management — Insertion of venous catheter under ultrasound guidance
  Other Names: management of catheter
Other: Cytology Specimen Collection Procedure — Collection of blood samples
  Other Names: Cytologic Sampling
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies the impact of radical cystectomy (surgery) on the expulsion (release) of circulating tumor cells into the blood stream in patients with bladder cancer. Significant surgery such as radical cystectomy may cause the expulsion of tumor cells. Studying the release of tumor cells into the circulation may help doctors understand the impact that radical cystectomy has on tumor metastasis and/or tumor recurrence.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To detect the numbers of circulating tumor cells (CTCs) during and following radical cystectomy in both the peripheral and central line.

SECONDARY OBJECTIVES:

I. To ensure the safety and of using the femoral vein to access the central venous blood supply for patients with primary bladder cancer and the withdrawal of blood from both a peripheral and central line.

OUTLINE:

Patients undergo placement of a central line via the right femoral vein and undergo open radical cystectomy (ORC). Blood samples are collected and analyzed for CTCs pre-surgery, at 30 minutes and 1 hour once ORC begins, post-surgery, and 7 days after surgery.

After completion of study, patients are followed up at 2 weeks and at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Must meet all inclusion and exclusion criteria
* Presence of a muscle invasive bladder tumor(s) (T2), specific for transitional cell carcinoma on pre-operative histology (i.e. biopsy or trans-urethral resection of bladder tumor [TURBT])
* Presence of a single bladder tumor lesion
* Patients are scheduled to undergo ORC at our institution
* Subjects must have given written informed consent to agree to participate
* Previous chemotherapy, and/or biological therapy for cancer are permitted provided that the acoustic properties of the tumor were not affected, but the subject should have recovered from the effects of these or of any prior surgery
* Subjects must be free of any clinically significant disease other than cancer that would interfere with the study evaluations
* Absolute neutrophil count (ANC) >= 1500 mm^-3
* Platelet count >= 100,000 mm^-3
* Hemoglobin >= 10 g/dl
* Prothrombin time (PT) =< 1.5 times upper limit of laboratory normal (ULN)
* Activated partial thromboplastin time =< 1.5 times ULN
* Total bilirubin < 1.5 times ULN
* Aspartate aminotransferase (AST) =< 3 times ULN
* Alkaline phosphatase < 2 times ULN, unless arising from bone

Exclusion Criteria:

* Subjects deemed unsuitable candidates and not medically optimized for ORC
* Subjects with tumors lying < 1 cm from sensitive structures such as the ureter, prostate or adjacent bowel
* Patients with presence of multiple bladder lesions
* Patients with pre-operative histologic confirmation of a bladder lesion other than transitional cell carcinoma
* Subjects on concurrent anticoagulant, or immunosuppressive medication
* Subjects on anti-cancer medication whether biologic or pharmaceutical
* Women who are pregnant or nursing (pregnancy test to be performed within 24 hours prior to high intensity frequency ultrasound [HIFU] treatment)
* Subjects assessed by consultant anesthetist as unsuitable for general anesthetic
* Absolute Contraindications: venous injury at the level of the femoral veins or proximally; known or suspected thrombosis of the femoral or iliac veins on the proposed side of venous annulation, ambulatory patient
* Relative Contraindications: presence of bleeding disorders; distortion of anatomy due to local injury or deformity; previous long-term venous catheterization; history of vasculitis; previous injection of sclerosis agents; previous radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with transitional cell bladder cancer scheduled to undergo open radical cystectomy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-02-05 (Estimated); Primary Completion 2019-02-05 (Estimated); Study Completion 2019-03-05 (Estimated)

PRIMARY OUTCOMES:
Number of CTCs in the blood drawn from central line | Up to post-operative day 7
  Will estimate the mean and standard deviation (possibly after log transformation to render data compatible with the assumptions of the normal distribution) at each time point (during and after radical cystectomy) as well as the changes over time.
Number of CTCs in the blood drawn from peripheral line | Up to post-operative day 7
  Will estimate the mean and standard deviation (possibly after log transformation to render data compatible with the assumptions of the normal distribution) at each time point (during and after radical cystectomy) as well as the changes over time.

SECONDARY OUTCOMES:
Incidence of complications during the cannulation of the femoral vein | Up to 1 month from discharge
  All complications will be recorded that occur during the insertion of femoral line, at any time during the surgical procedure or within 30 days of discharge from the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Inderbir Gill, MD, Principal Investigator — University of Southern California